CLINICAL TRIAL: NCT02151201
Title: Impact of Video Education on Influenza Vaccination Rate in Pregnancy
Brief Title: Impact of Influenza Vaccination in Pregnancy Video Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kenneth Goodman, MD, Staff Physician, Department of Family Medicine, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 13-1157
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Influenza
Keywords: pregnancy vaccination influenza education
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccination video education (Experimental): Influenza vaccination video education
  Interventions: Behavioral: Influenza vaccination video education
- Hand Washing video education (Placebo Comparator): Hand Washing vaccination video education
  Interventions: Behavioral: Hand washing video education

INTERVENTIONS:
Behavioral: Influenza vaccination video education — Influenza vaccination video education
  Arms: Influenza vaccination video education
Behavioral: Hand washing video education — Hand washing video education
  Arms: Hand Washing video education

SUMMARY:
We evaluated the impact of viewing an educational video about influenza vaccination in pregnancy just prior to a routine prenatal visit on vaccination health beliefs and vaccination rate. We hypothesized that the video would positively impact both vaccination health beliefs and vaccination rate compared to a control video.

DETAILED DESCRIPTION:
We studied the impact of influenza in pregnancy video education that was developed by the CDC and currently available to the public on the internet. We looked to see if viewing the video just prior to a routine scheduled prenatal visit could positively influence health beliefs regarding vaccination and improve the rate of vaccination that day. Patients were randomized to view the intervention video or a control video of similar length about hand washing. Pre visit and post visit questionnaires were given about vaccination health beliefs. We also asked if the shot had been recommended by the physician. One month after the visit, we used a structured phone interview to gather additional information regarding why participants who had not been vaccinated made that choice.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* English as primary language
* scheduled for a routine prenatal visit
* no documented influenza vaccination 2013-2014

Exclusion Criteria:

* Cleveland Clinic Employee
* high risk pregnancy
* allergy to eggs
* allergy to influenza vaccination

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Influenza Vaccination Rate | day of the prenatal visit
  The electronic medical record was used to establish if patients were vaccinated the day of their prenatal visit.

SECONDARY OUTCOMES:
Influenza Vaccination in Pregnancy Health Beliefs | day of the prenatal visit
Influenza vaccination in pregnancy health beliefs | Day of the appointment
  health beliefs regarding vaccination were tested on a 5 point likert-type scale before the video intervention and after the prenatal visit.

OTHER OUTCOMES:
Provider recommendation to become vaccinated | day of the appointment
  the post visit survey asked participants to recall if their physician had recommended that they get the flu shot that visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Goodman, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States